CLINICAL TRIAL: NCT01712373
Title: Study of Ginseng in Treatment of Fatigue in Multiple Sclerosis
Brief Title: Ginseng in Treatment of Fatigue in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Shemshaki, research assistant, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1270
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Fatigue
Keywords: Multiple sclerosis; Ginseng; Fatigue; Quality of life
MeSH Terms: conditions — Fatigue; Multiple Sclerosis | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginseng (Active Comparator): Ginseng, tablet, 250 mg, twice, 3 months
  Interventions: Drug: Ginseng
- Placebo (Placebo Comparator): Placebo, tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginseng — it is kind of drug
  Arms: Ginseng
Drug: Placebo — it is placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of Ginseng in treatment of fatigue and Quality of Life of MS patients.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is one of the most common non-traumatic causes of disability in the world. It is a chronic inflammatory and demyelinating disorder of the Central Nervous System (CNS) which affects individuals in the productive ages and causes a large burden for years to come. Fatigue is a common complaint and one of the least understood symptoms of MS

ELIGIBILITY:
Inclusion Criteria:

* definite diagnosis of relapsing-remitting MS (RRMS) by the MacDonald criteria with a baseline of Expanded Disability Status Score (EDSS)of less than 5.0

Exclusion Criteria:

* prior use of ginseng or any other tonic agents, glucocorticoids, warfarin, digoxin, aspirin, furosemide, caffeine, ephedra and anti-platelet agents within one month prior to enrollment;
* Pregnancy or lactation;
* history of renal failure; and,
* lack of appropriate adherence to the study protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Fatigue | at 3 months after treatment
  Modified Fatigue Impact Scale (MFIS)is a21-item (score range of each item: 0-4) questionnaire with the total score computed from 0 (no impact of fatigue) to 84 (maximum impact of fatigue) in three subscales containing: physical (9 items), cognitive (10 items) and psychosocial (2 items) aspects.

SECONDARY OUTCOMES:
Quality Of Life | at 3 months after treatment
  Quality Of Life Questionnaire (MSQOL-54) consisted of 54 questions (items), each one, assigned to a score ranging from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: mahboobe esfahani, MD, Principal Investigator — MD, Research Assistant
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran